CLINICAL TRIAL: NCT03167372
Title: Comparison of N-of-1 Trials of Light Therapy for Depressive Symptoms in Cancer Survivors
Brief Title: Pilot Comparison of N-of-1 Trials of Light Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ian Kronish, Associate Professor of Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAR1273; HHSN261200800001E (Other Grant/Funding Number: National Cancer Institute)
Record Dates: First submitted 2017-05-24; First posted 2017-05-30 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Cancer; Health Behavior; Depression
Keywords: Light Therapy; N-of-1
MeSH Terms: conditions — Neoplasms; Health Behavior; Depression

STUDY DESIGN:
Intervention Model Description: This study aims to assess the feasibility of conducting a randomized trial comparing two N-of-1 trials of light therapy in cancer survivors with depressive symptoms. In the first N-of-1 trial, participants will compare bright white light with dim red light therapy. In the second N-of-1 trial, participants will compare dim white light with dim red light. Participants will be randomized in a 2:1 ratio to either the N-of-1 bright white light vs dim red light experimental arm (N=20) or to a dim white vs dim red light therapy active comparator (N=10).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bright white light vs dim red light (Experimental): A balanced sequence (ABBA) over a 12 week period of bright white light and dim red light; alternating bright white and dim red light every 3 weeks.
  Subjects will receive 2 Litebook® Advantage lightboxes - 1 bright white and 1 dim red. Information such as mood, fatigue, sleep and light therapy side effects will be self-reported using a smartphone diary; physical activity and sleep will also be reported using a Fitbit Flex2 TM. Data visualization at 12 weeks.
  Interventions: Other: Litebook® Advantage; Other: Fitbit Flex2 TM
- Dim white light vs dim red light (Active Comparator): A balanced sequence (ABBA) over a 12 week period of dim white light and dim red light; alternating dim white and dim red light every 3 weeks.
  Subjects will receive 2 Litebook® Advantage lightboxes - 1 dim white and 1 dim red. Information such as mood, fatigue, sleep and light therapy side effects will be self-reported using a smartphone diary; physical activity and sleep will also be reported using a Fitbit Flex2 TM. Data visualization at 12 weeks.
  Interventions: Other: Litebook® Advantage; Other: Fitbit Flex2 TM

INTERVENTIONS:
Other: Litebook® Advantage — Standard system light therapy device used in an investigation to assess the feasibility of conducting a randomized trial design. The lightbox produces different wavelengths of the light identical to the peak wavelengths of the sun - bright white, dim white and red light.
  Other Names: Litebook Advantage Portable Light Therapy
Other: Fitbit Flex2 TM — Standard system activity and sleep tracker
  Other Names: Fitbit actigraph

SUMMARY:
This study compares the effect of two N-of-1 trials on study compliance with an N-of-1 protocol and on satisfaction with participation in an N-of-1 trial. Using within-person analyses, the study also compares the effect of different types of light therapy on mood, fatigue, sleep, physical activity, and side effects within a mild to moderately depressed cancer survivor population. Ten participants will be randomized to the bright white versus dim red light therapy N-of-1 trial, while the remaining 5 participants will be randomized to a dim white versus dim red light comparator N-of-1 trial.

DETAILED DESCRIPTION:
Fatigue or low energy levels, trouble sleeping and feeling down are symptoms that represent some of the most important concerns in cancer survivors, across a range of cancer types. Despite the impact of these symptoms on quality of life, previous studies have shown that few cancer survivors are receiving adequate treatment for these symptoms.

Light therapy involves the use of a light box (a box that lights up) in close proximity for a specified amount of time each day. There can be big differences in the way light therapy affects individual patients. Patients can learn whether this therapy is helpful to them by engaging in an N-of-1 trial. An N-of-1 trial is an experiment conducted with one individual (N refers to "number of individuals in the trial"). In an N-of-1 trial of light therapy, a patient can try light therapy to learn whether it is beneficial to them. All participants will receive two light boxes. The boxes will be labeled "A" and "B." Each light box will emit a different intensity of light. An app will send reminder notifications to participants' smartphones each morning to remind them which light box they should be using, depending on the week. They will be asked to use Box A or Box B each morning for 30 minutes per day for 12 weeks

The purpose of this study is to empower cancer survivors with symptoms of fatigue, trouble sleeping or who are feeling down to learn whether light therapy is helpful for them.

ELIGIBILITY:
Inclusion Criteria:

* History of cancer (not including basal cell or squamous cell carcinoma, or carcinoma in situ)
* Current mild to moderate severity depressive symptoms (PHQ-8 score 5 to 19)
* iPhone user

Exclusion Criteria:

* Has not completed primary cancer treatment including initial chemotherapy, surgical resection, or radiation therapy
* Non-English speaking
* Severe depression (PHQ-8 score >=20) or active suicidal ideations
* Other severe mental illness that would preclude participation in a study that requires extensive self-monitoring, including depression with psychotic features, other psychotic disorder, bipolar disorder, severe personality disorder
* <6 months life expectancy due to cancer or other severe medical illness
* Other severe medical illness that would preclude ability to do daily self-tracking
* Unavailable for follow-up over the course of the 3 month trial

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Protocol Compliance | Length of study (3 months)
  The proportion of participants randomized to the N-of-1 trial group who are compliant with the N-of-1 trial protocol
Participant Satisfaction | Length of study (3 months)
  The proportion of participants randomized to the N-of-1 trial who are satisfied with the N-of-1 trial protocol

SECONDARY OUTCOMES:
Depressive symptoms | Length of study (3 months)
  At the single-patient level in the bright white light experimental arm, effect of bright light versus dim white light on mood as measured by a daily visual analog scale.
Fatigue | Length of study (3 months)
  At the single-patient level in the bright white light experimental arm, effect of bright light versus dim white light on fatigue as measured by a daily visual analog scale.
Side effects | Length of study (3 months)
  At the single-patient level in the bright white light experimental arm, effect of bright light versus dim white light on days with perceived side-effects as measured by a smart phone daily diary.
Physical activity | Length of study (3 months)
  At the single-patient level in the bright white light experimental arm, effect of bright light versus dim white light on physical activity as measured by a Fitbit.
Treatment preference for bright white light therapy | Length of study (3 months)
  Within the bright white light experimental arm, the proportion who preferred to continue bright white light after the conclusion of the N-of-1 trial.

CONTACTS AND LOCATIONS:
Overall Officials: Ian Kronish, MD, MPH, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No